CLINICAL TRIAL: NCT00722917
Title: A Phase II, Randomized, Double-Blind, Placebo-and Active-Controlled, Multi-center Study to Determine the Efficacy and Safety of TAK-379 in Subjects With Type 2 Diabetes
Brief Title: Efficacy and Safety of TAK-379 in Adult Subjects With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Animal Toxicity Findings
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-379_201; U1111-1125-0948 (Registry Identifier: WHO)
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- TAK-379 25 mg QD (Experimental)
  Interventions: Drug: TAK-379
- TAK-379 100 mg QD (Experimental)
  Interventions: Drug: TAK-379
- TAK-379 200 mg QD (Experimental)
  Interventions: Drug: TAK-379
- Pioglitazone 30 mg QD (Active Comparator)
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-379 — TAK-379 25 mg, tablets, orally, once daily and pioglitazone placebo-matching tablets, orally, once daily for up to 12 weeks
  Other Names: Actos
  Arms: TAK-379 25 mg QD
Drug: TAK-379 — TAK-379 100 mg, tablets, orally, once daily and pioglitazone placebo-matching tablets, orally, once daily for up to 12 weeks
  Other Names: Actos
  Arms: TAK-379 100 mg QD
Drug: TAK-379 — TAK-379 200 mg, tablets, orally, once daily and pioglitazone placebo-matching tablets, orally, once daily for up to 12 weeks
  Other Names: Actos
  Arms: TAK-379 200 mg QD
Drug: Pioglitazone — Pioglitazone 30 mg, tablets, orally, once daily and TAK-379 placebo-matching tablets, orally, once daily for up to 12 weeks
  Other Names: Actos; AD4833
  Arms: Pioglitazone 30 mg QD
Drug: Placebo — TAK-379 placebo-matching tablets, orally, and pioglitazone placebo-matching tablets, orally, once daily for up to 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of multiple doses of TAK-379, once daily (QD), in subjects with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Type 2 diabetes is a metabolic disease that has reached epidemic proportions. The global incidence of this disease is estimated to increase from 120 million individuals to over 200 million by the year 2010. In type 2 diabetes, multiple metabolic defects contribute to hyperglycemia. These include insulin resistance, inadequate insulin secretion, and excessive hepatic glucose production. Nine classes of antihyperglycemic agents are currently approved for the treatment of type 2 diabetes (insulin, sulfonylureas, biguanides, alpha-glycosidase inhibitors, thiazolidinediones, glinides, glucagon-like peptide analogues, amylin analogues, and dipeptidyl peptidase 4 inhibitors). Each class acts by a unique mechanism on 1 or more of the metabolic defects.

Takeda Pharmaceutical Company Limited is developing TAK-379, a non-thiazolidinedione partial proliferator-activated receptor agonist for the treatment of type 2 diabetes mellitus. Study participation is anticipated to be approximately 4.5 months.

ELIGIBILITY:
Inclusion Criteria

* Historical diagnosis of type 2 diabetes mellitus without the chronic use of antidiabetic therapy and an 8 week history of diet and exercise.
* Historical diagnosis of type 2 diabetes mellitus on a stable dose of metformin as mono-therapy for at least 3 months prior to screening.
* Glycosylated hemoglobin between 7.5% and 10.0%, inclusive.
* Fasting C-peptide concentration is greater than or equal to 0.8 ng per mL.
* Any other chronic medications which have been stable for at least 4 weeks prior to Screening.
* Body mass index at Screening is greater than or equal to 23 kg/m2 and less than 45 kg/m2.
* Able and willing to monitor his or her own blood glucose concentrations with a home glucose monitor.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Compliance with single-blinded study medication during the run-in phase is at least 75% and does not exceed 125% based on tablet counts performed by the study staff.

Exclusion Criteria

* Systolic blood pressure is greater than 160 mm Hg, or diastolic pressure is greater than 100 mm Hg at repeat measurements.
* Any history of bladder cancer or has a history of cancer that has been in remission for less than 5 years prior to Screening (a history of basal cell carcinoma or Stage 1 squamous cell carcinoma of the skin is allowed).
* Glycosylated hemoglobin is less than 7.5% and greater than 10.0%.
* Creatine phosphokinase is greater than or equal to 5 times the upper limit of normal at screening.
* Hemoglobin is less than or equal to 12 g per dL for males and less than or equal to 10 g per dL for females.
* Alanine aminotransferase and aspartate aminotransferase are greater than or equal to 2.5 upper limit of normal.
* Total bilirubin is greater than or equal to 1.5 times the upper limit of normal at screening.
* Serum triglyceride concentration is greater than or equal to 400 mg per dL.
* Estimated glomerular filtration rate is less than or equal to 60 mL per min using the Modification of Diet in Renal Disease equation or the Cockroft-Gault equation.
* Abnormal thyroid-stimulating hormone as defined by central laboratory normals.
* Positive test result for hepatitis B surface antigen or hepatitis C antibody.
* Urine albumin to creatinine ratio is greater than or equal to 1000 μg per mg at screening.
* History of microscopic or macroscopic hematuria.
* Two consecutive unexplained positive urinalysis dip-stick and greater than or equal to 3 red blood cells per high-powered field on two consecutive measurements.
* History of laser treatment for proliferative diabetic retinopathy within 6 months prior to Screening.
* Diabetic gastroparesis that in the investigator's opinion is moderate or severe and hence may impair absorption of study medication.
* The subject has New York Heart Association Class III or IV heart failure.
* Has had coronary angioplasty, coronary stent placement, coronary bypass surgery, myocardial infarction, unstable angina pectoris, clinically significant abnormal electrocardiogram, cerebrovascular accident or transient ischemic attack within 6 months prior or at Screening.
* History of any hemoglobinopathy that may affect determination of glycosylated hemoglobin.
* Received treatment with probucol within 1 year of randomization.
* Donated or received any blood products within 12 weeks prior to Screening.
* Received treatment for greater than 7 days within 8 weeks prior to randomization or is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * oral or systemically injected glucocorticoids
  * Prescription or over the counter weight-loss drugs
  * Peroxisome proliferator-activated receptor agonists, including fibric acid derivatives
  * Niacin
  * Ezetemibe
  * Bile-acid binding agents
  * warfarin
  * phenytoin
  * any alteration in lipid-lowering medication (change in dosage or drug)
* Chronically treated with insulin.
* Received any investigation drug within 4 weeks prior to Screening.
* History of infection with hepatitis B, hepatitis C, or human immunodeficiency virus.
* Hypersensitive to TAK-379 or its excipients.
* History of drug abuse or a history of alcohol abuse within 2 years prior to Screening.
* Any other physical or psychiatric disease or condition that in the judgment of the investigator may affect life expectancy or may make it difficult to successfully manage and follow the subject according to the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Glycosylated Hemoglobin | Week 12 or Final Visit

SECONDARY OUTCOMES:
Change from baseline in glycosylated hemoglobin. | Weeks 4 and 8 or Final Visit
Change from baseline in fasting plasma glucose. | Weeks 1, 2, 4, 8 and 12 or Final Visit
Change from baseline in body weight. | Weeks 4, 8 and 12 or Final Visit
Number of patients with elevation of alanine aminotransferase greater than three times the Upper Limit of Normal during treatment. | Week 12 or Final Visit
Plasma concentrations of TAK-379 and its metabolite M-I via a sparse sampling population approach. | Week 12 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (8):
- United States (8):
  - Artesia, California
  - Norwalk, California
  - Santa Ana, California
  - Santa Monica, California
  - Panama City, Florida
  - Cranston, Rhode Island
  - Dallas, Texas
  - Houston, Texas